CLINICAL TRIAL: NCT00287170
Title: Pilot, Open-Label, Randomized, Parallel Group Study to Evaluate Clinical/ and Immunological Efficacy/Safety of Locally Delivered 6-MP or Calcitriol vs Purinethol in Non-Steroid Dependent Patients With Active CD
Brief Title: Efficacy Study of Targeted, Local Delivery of Drugs to Treat Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva GTC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2/13/6MP:CAL-01
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Local Ileal Delivery; Delayed-Release Formulations; 6-Mercaptopurine; Calcitriol
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Drug: Delayed Release 6MP or Calcitriol vs. Purinethol

SUMMARY:
The study is being undertaken to evaluate whether delayed-release medications, designed to begin to open in the lower intestinal tract, the main site of Crohn's Disease, are more effective than standard systemically delivered drugs to promote remission or response in CD patients. It is hypothesized that the delayed-release medications will go right to the injured tissue and heal the disease more quickly.

The delayed-release test drugs are 6-mercaptopurine (at a dose of 40 mg daily) or calcitriol (at a dose of 5 mcg three times a week) versus Purinethol (6-MP at a dose of 1-2 mg/kg body weight daily). Calcitriol is a synthetically manufactured replica of a natural substance in the body that is derived from Vitamin D. There is much medical evidence that shows that lack of Vitamin D can be a possible risk factor in developing autoimmune disorders, including Crohn's Disease. Moreover, calcitriol has been shown in animal models to improve the symptoms of Crohn's Disease.

DETAILED DESCRIPTION:
This pilot clinical study is designed to evaluate the efficacy and safety of oral administration of novel, delayed-release test formulations, for targeted delivery to the ileum in Crohn's Disease patients. The local delivery drugs (delayed-release formulations of 6-mercaptopurine or calcitriol) will be compared to standard Purinethol treatment after 12 weeks of treatment to evaluate:

* (1) local intestinal mucosal inflammation and damage as shown by markers of biopsy tissue (CDEIS and pathologist review of biopsies);
* (2) Clinical symptoms of active Crohn's Disease [CDAI scores- remission <150; response- a drop of 100 points from baseline; IBDQ scores- >= 180 indicative of remission]; and
* (3)Systemic improvement as shown by blood immunological and inflammatory markers (CRP and ESR).

It is hypothesized that since CD is a localized autoimmune inflammation of the intestinal mucosa, a far more effective, and potentially safer treatment would be targeted, local delivery of effective drugs directly to the disease site. The drug would be concentrated in the specific area of disease, while unwanted systemic side effects would be minimized. The drugs selected for evaluation are 6-MP (a mainstay of CD treatment for over 30 years) and calcitriol, a synthetically manufactured Vitamin D derivative, which is being evaluated in many studies for its impressive immunomodulatory effects in cancer, MS and other autoimmune disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients, aged 18-75 years with moderate Crohn's Disease (CDAI score >=220 and <=400 at screening), with or without adjunctive mesalamine treatment, 12 with involvement of the ileum and three without ileal involvement
* Definitive diagnosis of active inflammatory CD with fibrostenosing and/or fistulizing/perforating CD types ruled out based on clinical and radiological or endoscopic or pathological findings, within the previous 6 months

Exclusion Criteria:

* Body weight below 42.5 kg
* Subjects who have received either methotrexate, cyclosporine or anti-TNFalpha (infliximab, Remicade), anti-integrin (namixilab) in the past 3 months
* Subjects who are taking allopurinol, sulfasalazine, valerian, warfarin and corticosteroids,including budesonide and prednisone within 28 days prior to and throughout the study
* Previous bowel resection, including prior colostomy, ileostomy or colectomy with ileorectal anastomosis
* Symptomatic stenosis or ileal strictures; x-ray evidence of fibrosed bowel
* Subjects with ulcerative colitis or short bowel syndrome
* Subjects who present with, or with a history of persistent intestinal obstruction, bowel perforation, uncontrolled GI bleed or abdominal abscess or infection, toxic megacolon
* Subjects with fistulizing CD or isolated small bowel CD
* Subjects with evidence of other serious infectious, autoimmune, hepatic,nephritic or systemic disease or compromised organ function
* Subjects with a history of GI tract malignancy or IBD-associated malignant changes in the intestines

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-07; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Remission-defined as a CDAI (Crohn's Disease Activity Index) of <150 | 12 weeks
Response- defined as a fall in the CDAI by 100 points or more from baseline | 12 weeks

SECONDARY OUTCOMES:
Improvement in ESR (Erythrocyte Sedimentation Rate), CRP (C-Reactive Protein) levels, and IBDQ (Inflammatory Bowel Disease Questionnaire) >=180 indicative of remission

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel